CLINICAL TRIAL: NCT07238374
Title: The Effect of Various Music Therapies and Robotic Parrot Therapy on Anxiety and Fatigue Levels in Hemodialysis Patients: A Randomized Controlled Study
Brief Title: The Effect of Various Music Therapies and Robotic Parrot Therapy on Anxiety and Fatigue Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Asst. Prof., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCS04082023
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Renal Failure Chronic; Anxiety; Fatigue
Keywords: Anxiety; Complementary therapies; Fatigue; Hemodialysis; Music therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anxiety Disorders; Fatigue | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: The sample size was calculated using the G*Power 3.1.9.6 program with an error rate of α=0.05. Since there were no previous four-group studies on the subject, no reference could be used. with an effect size of 0.2 and a target test power of 0.80 (90%), a total of 68 patients (17 per group) were calculated for the four groups (music-repeating robotic parrot, live music, live ney sound, and control group). Taking into account situations such as wanting to leave the study or death during the research, each group was increased by 10%, and a total of 76 patients were included in the study, with 19 patients in each group. The study was completed with 64 HD patients.
Who Masked: Investigator
Masking Description: After explaining the purpose of the study and completing the consent forms, the researcher conducted a double-blind randomized controlled clinical trial to reduce bias. In this context, the two researchers who applied the data collection tools and the third researcher who analyzed the data were not informed about which experimental groups (music-repeating robotic parrot, live music, live ney sound) or control group the hemodialysis patients were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Music-Repeating Robotic Parrot (Experimental): Before the study (week 0/pre-test), data were collected from all participants using the "Patient Information Form", "Fatigue Severity Scale" and "Beck Anxiety Scale". The "Fatigue Severity Scale" and "Beck Anxiety Scale" were re-administered at the end of the 1st and 2nd months of the therapy process. Following the end of the application, patients were monitored without therapy for 8 weeks, and these scales (Fatigue Severity Scale and Beck Anxiety Scale) were evaluated for the last time in the 3rd and 4th months (16th week/final test).
  Interventions: Other: Music-Repeating Robotic Parrot (Pet therapy)
- Live Music (Experimental): Before the study (week 0/pre-test), data were collected from all participants using the "Patient Information Form", "Fatigue Severity Scale" and "Beck Anxiety Scale". The "Fatigue Severity Scale" and "Beck Anxiety Scale" were re-administered at the end of the 1st and 2nd months of the therapy process. Following the end of the application, patients were monitored without therapy for 8 weeks, and these scales (Fatigue Severity Scale and Beck Anxiety Scale) were evaluated for the last time in the 3rd and 4th months (16th week/final test).
  Interventions: Other: Live Music (Pet therapy)
- Live Ney Sound (Experimental): Before the study (week 0/pre-test), data were collected from all participants using the "Patient Information Form", "Fatigue Severity Scale" and "Beck Anxiety Scale". The "Fatigue Severity Scale" and "Beck Anxiety Scale" were re-administered at the end of the 1st and 2nd months of the therapy process. Following the end of the application, patients were monitored without therapy for 8 weeks, and these scales (Fatigue Severity Scale and Beck Anxiety Scale) were evaluated for the last time in the 3rd and 4th months (16th week/final test).
  Interventions: Other: Live Ney Sound (Pet therapy)
- Control Group (No Intervention): Patients in this group did not receive any intervention from the researcher for 16 weeks. The "Patient Information Form," "Fatigue Severity Scale" and "Beck Anxiety Scale" were administered at the pre-test. Subsequently,"Fatigue Severity Scale" and "Beck Anxiety Scale" measurements were repeated in the 1st, 2nd, 3rd, and 4th months (16th week/final test).

INTERVENTIONS:
Other: Music-Repeating Robotic Parrot (Pet therapy) — Patients in the experimental groups underwent 30-minute therapy sessions 3 days a week for 8 weeks. In robotic parrot therapy, patients were asked to sing and listen to the robotic parrot's repetition.
  Arms: Music-Repeating Robotic Parrot
Other: Live Music (Pet therapy) — Patients in the experimental groups underwent 30-minute therapy sessions 3 days a week for 8 weeks. In live music therapy, songs were performed accompanied by instruments such as guitar and darbuka.
  Arms: Live Music
Other: Live Ney Sound (Pet therapy) — Patients in the experimental groups underwent 30-minute therapy sessions 3 days a week for 8 weeks. In live ney sound therapy, only instrumental music was performed using the ney.
  Arms: Live Ney Sound

SUMMARY:
This study aimed to evaluate the effect of robotic parrot therapy, live music, and live ney sound therapy on anxiety and fatigue levels in hemodialysis patients.

DETAILED DESCRIPTION:
Although the life-saving effects of hemodialysis treatment are indisputable, this treatment process can also bring serious problems. In particular, the frequency and length of hemodialysis sessions, inherent in their nature, cause physical exhaustion in patients and also create a significant psychological burden. Clinical studies and observational research have demonstrated that high levels of anxiety and persistent fatigue are frequently observed in patients undergoing hemodialysis. The prevalence of these symptoms is a consistent finding that negatively affects both patients' overall quality of life and their adherence to the treatment regimen. In this context, in addition to standard medical treatment approaches, the need for holistic and non-pharmacological support methods focused on supporting patients' psychological well-being has become critically important.

In line with this need, complementary practices such as music therapy and pet therapy are gaining increasing attention in the field of chronic disease management. Music therapy has emerged as an effective tool in alleviating symptoms such as anxiety, depression, and pain in hemodialysis patients, as demonstrated by evidence-based studies. The positive effects of listening to instrumental music or music selected by the patient on psychological symptoms are also supported by meta-analyses. However, while the vast majority of studies in music therapy focus on passive listening, the effects of different instrumental types of live music, which may have a higher therapeutic effect, have not been sufficiently investigated. In particular, there are very few studies examining the specific and comparative interactions on the symptom of fatigue, which is common and difficult to treat in hemodialysis patients. Therefore, a deeper understanding of the mechanisms of action of different live music approaches is a primary research requirement.

On the other hand, pet therapy has been clearly proven to reduce anxiety and loneliness levels in studies conducted on the general population and psychiatric patients. Parrots, in particular, have been used in therapeutic work due to their social interaction and vocal mimicry abilities. In the reviewed literature, only one unpublished doctoral thesis has been found internationally that uses live parrot therapy in mental health. In Turkey, no studies using parrot therapy have been found. However, the introduction of live animals into environments with high infection risks, such as dialysis units, is not recommended due to practical and ethical barriers, including strict hygiene standards and allergy potential. These limiting factors create a need for robotic alternatives that can mimic the social interaction and distraction benefits of pet therapy.

In this context, robotic parrots are an innovative tool that can deliver the benefits of pet therapy without hygiene and safety concerns. Previous research has shown that parrot-inspired robots are successful in capturing the attention and increasing the social participation of individuals who experience difficulties in social interaction. Therefore, it is thought that the use of such interactive robotic parrots with sound and music repetition features during hemodialysis sessions could create a new source of emotional and cognitive support for patients and have a positive effect on symptoms such as anxiety and fatigue.

Considering all this information, this study aims to compare the effects of robotic parrot therapy and different instrumental live music therapy approaches on anxiety and fatigue in hemodialysis patients for the first time using a double-blind randomized controlled design. The scientific data obtained will guide the development of evidence-based and innovative intervention protocols that support traditional medical care .

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Receiving hemodialysis treatment 3 times per week,
* Having received regular hemodialysis treatment for at least 6 months,
* Being conscious and able to communicate, with no impairment in mental and cognitive functions,
* Not having previously received music therapy or pet therapy.

Exclusion Criteria:

* Refusal to participate in the study,
* Being 18 years of age or younger,
* Having severe hearing loss,
* Hemodynamic status not being stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 16 week
  The scale generally consists of 9 items. The items inquire about the effect of fatigue on cognitive functions such as motivation, exercise, physical functioning, daily living activities, and attention/concentration. The rating uses a 7-point Likert-type format. The individual indicates their level of agreement with each item by selecting a score between 1 (strongly disagree) and 7 (strongly agree). The total score ranges from 9 to 63. A total score of 36 or higher generally indicates the presence of clinically significant fatigue.
  Before the study (week 0/pre-test), data were collected from all participants using the "Fatigue Severity Scale". The Fatigue Severity Scale were re-administered at the end of the 1st and 2nd months of the therapy process. Following the end of the application, patients were monitored without therapy for 8 weeks, and these scale were evaluated for the last time in the 3rd and 4th months (16th week/final test).
Beck Anxiety Scale | 16 week
  The Scale measures both the cognitive/emotional and somatic (physical) components of anxiety, asking participants to rate the degree to which each symptom has bothered them in the past week on a scale from 0 (Not at all) to 3 (To a great extent). The total score obtained from the scale, ranging from 0 to 63, reflects the severity of anxiety; according to common interpretation, a score between 8 and 15 indicates mild anxiety, between 16 and 25 indicates moderate anxiety, and between 26 and 63 indicates severe anxiety.
  Before the study (week 0/pre-test), data were collected from all participants using the "Beck Anxiety Scale". TheBeck Anxiety Scale were re-administered at the end of the 1st and 2nd months of the therapy process. Following the end of the application, patients were monitored without therapy for 8 weeks, and these scale were evaluated for the last time in the 3rd and 4th months (16th week/final test).

CONTACTS AND LOCATIONS:
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll decide later